CLINICAL TRIAL: NCT01637714
Title: The Effects of Multi-strain Probiotics in Adults With Diarrhea Predominant Irritable Bowel Syndrome: Double-blind, Randomized, Placebo-controlled Trial
Brief Title: The Effects of Multi-strain Probiotics in Adults With Diarrhea Predominant Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Probiotics for IBS
Record Dates: First submitted 2012-06-21; First posted 2012-07-11 (Estimated); Last update posted 2013-06-18 (Estimated); Status verified 2013-06

CONDITIONS: Diarrhea Predominant Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Multi-strain probiotics (Experimental)
  Interventions: Drug: Multi-strain probiotics
- Placebo powder (Placebo Comparator)
  Interventions: Drug: Placebo powder

INTERVENTIONS:
Drug: Multi-strain probiotics — * B. longum BORI: 1 x 109
  * B. bifidum BGN4: 1 x 109
  * B. lactis AD011: 1 x 109
  * B. infantis IBS007: 1 x 109
  * Lactobacillus acidophilus AD031: 1 x 109
  three times a day, within 10 minutes after meal, per oral with water
  Arms: Multi-strain probiotics
Drug: Placebo powder — same taste, shape, dosage as experimental drug
  three times a day, within 10 minutes after meal, per oral with water
  Arms: Placebo powder

SUMMARY:
The investigators will evaluate the efficacy of multi-strain probiotics in adults with diarrhea predominant irritable bowel syndrome.

ELIGIBILITY:
Inclusion Criteria:

* willing to consent/undergo necessary procedures
* between the age of 19 and 75 years
* diarrhea predominant irritable bowel syndrome (satisfied with Rome II criteria)

Exclusion Criteria:

* uncontrolled hypertension (Blood pressure > 180/110 mmHg)
* uncontrolled diabetes mellitus (FBS > 200 mg/dL)
* malignancy, cerebrovascular disease, cardiovascular disease
* history of abdominal surgery except appendectomy and hernia repair
* inflammatory bowel disease
* clinically or laboratory-confirmed gastroenteritis
* the use of motility drug or dietary fiber supplement in 2 weeks
* serum Cr > 2 x Upper normal limit
* AST or ALT > 2 x Upper normal limit
* Pregnancy, Lactating woman

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
change of Irritable bowel syndrome symptom severity score (IBS-SSS) | after 8 weeks
  Severity and frequency of abdominal pain / abdominal bloating / bowel habitus / interfere degree of daily life

SECONDARY OUTCOMES:
Stool frequency and form | after 4 weeks and 8 weeks
  Stool frequency (greater than 3 bowel movements/day or less than 3 bowel movements/week) Stool form (lumpy / hard or loose / watery stool)
Symptom control of irritable bowel syndrome | after 4 weeks and 8 weeks
Improvement of overall symptom in patient with irritable bowel syndrome | after 4 weeks and 8 weeks
Assessment for quality of life related with irritable bowel syndrome | after 4 weeks and 8 weeks
Assessment for patient satisfaction after administration completion | after 4 weeks and 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Joo Sung Kim, M.D.,PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea